CLINICAL TRIAL: NCT07071051
Title: Exploring the Effect of Calaspargase Pegol on the Coagulation System in Pediatric Acute Lymphoblastic Leukemia (ALL) Patients: Pilot Study
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 24-012104; NCI-2025-04657 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-012104 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Childhood Acute Lymphoblastic Leukemia; Childhood Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo collection of blood samples and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates the impact of calaspargase pegol (Cal-PEG) on the coagulation system in pediatric patients with acute lymphoblastic leukemia/lymphoma (ALL).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the impact of Calaspargase Pegol (Cal-PEG) on the coagulation system in pediatric ALL patients.

II. Compare bleeding and thrombotic events associated with Cal-PEG to historical controls treated with pegaspargase.

OUTLINE: This is an observational study.

Patients undergo collection of blood samples and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-21.5 years
* Confirmed diagnosis of acute lymphoblastic leukemia/lymphoma
* Planned treatment with Cal-PEG
* Informed consent obtained from parents or guardians

Exclusion Criteria:

* Pre-existing coagulation disorders
* Known hypersensitivity to asparaginase products
* Liver failure
* Any acute or chronic disease that is known to affect coagulation testing (e.g. nephrotic syndrome)
* Currently pregnant

Ages: 2 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be pediatric patients diagnosed with ALL and scheduled to receive Cal-PEG as part of their treatment regimen.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in coagulation - frequency | Baseline (either before first dose or after at least 6 weeks from last Cal-PEG administration); approximately 4, 11, 18, and 39 days after Cal-PEG administration
  Frequency of coagulation changes in patients with Acute Lymphoblastic Leukemia (ALL) who receive Cal-peg as part of their treatment. Blood samples will be collected at baseline (pre-treatment: either before first dose or after at least 6 weeks from last Cal-PEG administration) and at 4-, 11-, 18-, and 39-- -days post-Cal-PEG administration (time points can be adjusted based on routine clinical testing within ± 4 days).
Change in coagulation - duration | Baseline (either before first dose or after at least 6 weeks from last Cal-PEG administration); approximately 4, 11, 18, and 39 days after Cal-PEG administration
  Duration of coagulation changes in patients with Acute Lymphoblastic Leukemia (ALL) who receive Cal-peg as part of their treatment. Blood samples will be collected at baseline (pre-treatment: either before first dose or after at least 6 weeks from last Cal-PEG administration) and at 4-, 11-, 18-, and 39-- -days post-Cal-PEG administration (time points can be adjusted based on routine clinical testing within ± 4 days).
Incidence of clinically relevant hematologic or thrombotic adverse events | Up to 12 weeks
  Assessed according to Common Terminology Criteria for Adverse Events (CTCAE) criteria. Will describe clinically relevant hematologic or thrombotic adverse events in patients with ALL who receive Cal-PEG as part of their treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine B. O'Keefe, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials